CLINICAL TRIAL: NCT00206934
Title: The Effects of Increased Central Serotonergic Activity on Psychophysiological Parameters of Human Information Processing
Brief Title: The Effects of Increased Central Serotonergic Activity on Information Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Lundbeck Foundation (Other); Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Birte Glenthoj, Professor of Psychopharmacology and Neuropsychiatry, Danish Center for Neuropsychiatric Schizophrenia Research
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 363037-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2008-07

CONDITIONS: Healthy Volunteers
Keywords: PPI; P50 suppression; P300; mismatch negativity; escitalopram
MeSH Terms: interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Escitalopram
- 2 (Placebo Comparator)
  Interventions: Drug: escitaolpram

INTERVENTIONS:
Drug: Escitalopram — Either 10 mg of escitalopram or placebo will be administered to a group of healthy volunteers
  Other Names: Cipralex
  Arms: 1
Drug: escitaolpram — Either 15 mg of escitalopram or placebo will be administered to healthy volunteers
  Other Names: Cipralex
  Arms: 2

SUMMARY:
It is of great clinical relevance to know if selective serotonin re-uptake inhibitors affect information processing. Our hypothesis was that aspects of information processing would be disturbed whereas others would improve.

DETAILED DESCRIPTION:
Numerous studies point to an increased serotoninergic activity in schizophrenia. Additionally, patients with schizophrenia often show reduced filtering of sensory information, which is reflected in reduced P50 suppression and reduced prepulse inhibition of the startle refex (PPI). Currently, the reports in literature on the effects of serotonergic agonists on sensory gating in humans are inconclusive. In an initial study performed in our laboratory, however, we found reduced P50 suppression following administration of imipramine (a combined serotonin- and noradrenalin reuptake inhibitor) to healthy volunteers. This result provides evidence for the involvement of either serotonergic, noradrenergic, or a combination of both pathways in sensory gating. In numerous animal studies however, sensory gating is reduced by agonists of 5-HT, which suggests a serotonergic, rather than a noradrenergic, involvement in sensory gating. Therefore, in a follow-up study, the effects of a selective serotonin reuptake inhibitor (escitalopram) will be investigated on sensory gating parameters of healthy volunteers. To further extend the data of our initial study, the subjects will additionally be tested for two more psychophysiological parameters of attention that are usually found to be disturbed in patients with schizophrenia, i.e. mismatch negativity and selective attention. The design will be a double blind, placebo controlled experiment, in which a single dose of escitalopram or placebo will be given to healthy, non-smoking male volunteers on two occasions, separated by at least a week, after which the subjects will be tested in the psychophysiological test battery.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* Good Physical and Mental Health meeting criteria "never mentally ill", which will be evaluated with a medical history checklist, ECG
* Non smokers

Exclusion Criteria:

* Current use of any medication
* Any subject who has received any investigational medication within 30 days prior to the start of this study
* History of neurologic illness
* History of psychiatric illness in first-degree relatives, evaluated with DSM-IV criteria
* History of alcohol and drug abuse. Positive urine screening for amphetamine, cocaine, cannabis, or esctacy.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2005-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The PPI (Prepulse Inhibition of the Startle Response) task | Once, 3.5 hrs after intake of capsule
The P50 Suppression task | Once, 3.5 hrs after intake of capsule
The P300 ERP task | Once, 3.5 hrs after intake of capsule
The mismatch negativity (MMN) task | Once, 3.5 hrs after intake of capsule

CONTACTS AND LOCATIONS:
Overall Officials: Birte Glenthoj, MD, DMSc., Study Director — Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychaitric Center Glostrup, Ndr. Ringvej, DK-2600 Glostrup, Denmark
Locations (1):
- Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychiatric Center Glostrup, Glostrup Municipality, Denmark

REFERENCES:
- See also: Center for Neuropsychiatric Schizophrenia Research (CNSR) — http://www.cnsr.dk